CLINICAL TRIAL: NCT04127591
Title: Differential Expression and Analysis of Peripheral Plasma Exosome miRNA in Patients With Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Bin He, M.D./Ph.D., Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-19-010
Record Dates: First submitted 2019-10-14; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- myocardial infarction group: Patients admitted with the diagnosis of myocardial infarction.
  Interventions: Other: exosome
- Blank control group: Patients admitted without the diagnosis of myocardial infarction.
  Interventions: Other: exosome

INTERVENTIONS:
Other: exosome — Collect exosomes in peripheral blood of patients and extract miRNAs from them.

SUMMARY:
The aim of this study is to determine the miRNA expression profile in peripheral blood exosomes of patients with myocardial infarction and to investigate its relationship with myocardial infarction.

DETAILED DESCRIPTION:
Collect exosomes in peripheral blood of patients with myocardial infarction, compare the expression of miRNA with healthy volunteers, find out the miRNAs with significant differences, and explore its relationship with the development of myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years ST elevation by ECG diagnostic of STEMI Evidency of coronary occlusion in coronariography Signed informed consent

Exclusion Criteria:

* Patients who will undergo immediate PCI Pregnant and lactating women Patients with mental disorders Patients are using other experimental drugs; Refusal to provide informed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-10-20 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Determination of differential expression of miRNA by second-generation sequencing technology | Day 7

SECONDARY OUTCOMES:
Diagnostic value of the differential microRNAs evaluate by qPCR in patients of myocardial infarction | Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided